Official Title: Management of Spontaneous Ruptured Hepatocellular Carcinoma

- Partial Hepatectomy and Prognosis: A Retrospective Study

**NCT number: Not available** 

Date of the document: 05/03/2018

## Statistical analysis plan

All of the analyses were carried out using SPSS 24.0 (IBM), and a two-sided P<0.05 was considered statistically significant.

- Univariate and multivariate analysis of the predictive factors associated with overall survival (OS) before PSM: surgery or non-surgical treatment is (or not) an independent risk factor of overall survival.

The variables included are: age, sex, tumor size, tumor number, MVI, cirrhosis, portal hypertension, treatment, hemorrhagic shock, distant metastasis, AST, AFP, platelet, hemoglobin, sorafenib, Child-Pugh grade.

Statistical analysis method: univariate analysis was performed using the Kaplan-Meier method compared by the log-rank test; multivariate analysis was performed using the COX regression model.

A comparison of the clinicopathologic characteristics of all of the patients between the
partial hepatectomy group and the non-surgical treatment group after PSM: there is no
significance for patients' characteristics after PSM.

The variables included in PSM are: age, sex, tumor size, tumor number, MVI, cirrhosis, portal hypertension, hemorrhagic shock, hemoglobin, red blood cell (RBC), transfusion during hospitalization, a-fetoprotein (AFP), aspartate aminotransferase (AST), albumin, total bilirubin.

Statistical analysis method: PSM, a caliper of 0.5, 0.3, 0.2, 0.1, 0.05, 0.02, 0.01 would be used.

Univariate and multivariate analysis of the predictive factors associated with OS after
 PSM: surgery or non-surgical treatment is (or not) an independent risk factor of overall
 survival.

The variables inclued are: age, sex, tumor size, tumor number, MVI, cirrhosis, portal hypertension, treatment, hemorrhagic shock, distant metastasis, AST, AFP, platelet, hemoglobin, Sorafenib, Child-Pugh grade.

Statistical analysis method: univariate analysis was performed using the Kaplan-Meier method compared by the log-rank test; multivariate analysis was performed using the

COX regression model.

 Comparison of OS and recurrence-free survival (RFS) between the emergency partial hepatectomy group and the staged partial hepatectomy group.

Statistical analysis method: univariate analysis was performed using the Kaplan-Meier method compared by the log-rank test.

6. Comparison of OS and RFS between the staged early partial hepatectomy group and the staged late partial hepatectomy group.

Statistical analysis method: univariate analysis was performed using the Kaplan-Meier method compared by the log-rank test.

7. Difference in 30-day mortality of peritoneal dissemination between the groups at different times.

Statistical analysis method: Pearson's  $\chi 2$  test,  $\chi 2$  test with Yates' correction and Fisher's exact test.

8. Univariate and multivariate logistic regression analysis of postoperative peritoneal dissemination.

The variables inclued are: age, sex, tumor size, tumor number, MVI, cirrhosis, estimated intraperitoneal bleeding, Child-Pugh grade, tumor differentiation, resection margin, type of hepatectomy, timing of hepatectomy.

Statistical analysis method: univariate and multivariate logistic regression analysis.